CLINICAL TRIAL: NCT03035669
Title: Effects of Mindfulness Training on Emotion Regulation and Social Cognition, a Psychophysiological and Neuroimaging Randomized Controled Study.
Brief Title: Effects of Mindfulness Training on Emotion Regulation and Social Cognition.
Acronym: MFN&SOCCOG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Humboldt-Universität zu Berlin (Other)
Collaborators: Comisión Nacional de Investigación Científica y Tecnológica (Other Government)
Responsible Party: Principal Investigator, Simon Guendelman, Medical doctor, doctorate candidate., Humboldt-Universität zu Berlin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HumboldtUB
Record Dates: First submitted 2016-11-30; First posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Stress, Psychological; Emotional Stress; Social Cognition; Mindfulness
MeSH Terms: conditions — Stress, Psychological | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness group (Experimental): Mindfulness based stress reduction: 8 week program, including meditation, body-awareness, and yoga practices. Daily assignments and home practices during 50 minutes per day.
  Interventions: Behavioral: Mindfulness group
- Reading group (Active Comparator): Reading and sharing group: 8 week program, including readings, interpersonal exchanges, group discussion, listening and role playing exercises. Daily assignments and home practices during 50 minutes per day.
  Interventions: Behavioral: Reading group

INTERVENTIONS:
Behavioral: Mindfulness group — 8 week program
  Other Names: mindfulness based stress reduction
  Arms: Mindfulness group
Behavioral: Reading group — 8 week program
  Other Names: Reading and sharing group
  Arms: Reading group

SUMMARY:
The present study will investigate the effects of a mindfulness training on emotion regulation and social cognition, using several psychological, behavioral, psychophysiological and neuroimaging methods.

DETAILED DESCRIPTION:
The aim of the present study is to evaluate the impact of a mindfulness intervention, particularly the mindfulness-based stress reduction (MBSR), on the capacities of emotion regulation and social cognition, in caring/helping professions which are vulnerable to stress. In the context of a longitudinal intervention study, a randomized controlled trial, the efficacy of the MBSR to increase the capacity for self-emotion regulation, empathic attunement, and compassion capacities will be measured. For doing this, several psychological, behavioral, psychophysiological and neuroimaging brain measurements will be used.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers: Men or women
* Right-handed
* Normal or corrected-to-normal visión
* German as a first language
* No history of neurological or psychiatric problems, or use of controlled medication that might interfere with emotion or attention.
* No symptoms of claustrophobia
* Written informed consent form to participate in the study and neuro-imaging experiment.

Exclusion Criteria:

* Chemical dependence, including nicotine and alcohol
* Dementia or psychotic condition.
* Depression or use of antidepressants
* Pregnant or breast-feeding women
* Prior MBSR class or regularly practicing mindfulness meditation (or yoga) for three or more months.
* Non-controlled severe medical disease that might interfere with the performance of the study, such as neoplasias, cardiopathies, digestive pathologies, diabetes mellitus type I or type II
* Neoplasias in the central nervous system
* Tremor or dystonia in cephalic segment that hinders the performance of the MRI study (tremor equal to or higher than 3 in each corporal segment, according to the UPDRS scale)
* Fulfillment of any criterion of contraindication for the MRI exam (for instance, metallic implants, claustrophobia, pregnancy, use of pacemaker; intracranial aneurism clip; cochlear implants).
* Presence of odontological devices that might disturb the magnetic field or any sources of variation of the magnetic susceptibility
* Any other conditions the investigator might deem problematic for the inclusion of the volunteer in a trial of this nature will also be considered.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Activation changes in emotions related brain regions. Measured by significant changes in the BOLD (blood oxygenated level dependent) signal from task based functional magnetic resonance imaging. | first acquisition period during 3 weeks before the intervention, second acquisition period during 3 weeks after the intervention.
Changes in resting state functional connectivity within brain networks. Measured by significant changes in intrinsic functional connectivity parameters, estimated from the resting state BOLD signal, during functional magnetic resonance imaging. | first acquisition period during 3 weeks before the intervention, second acquisition period during 3 weeks after the intervention.

SECONDARY OUTCOMES:
Changes in resting state functional connectivity between inter-networks connectivity. | first acquisition period during 3 weeks before the intervention, second acquisition period during 3 weeks after the intervention.
  Changes between brain networks connectivity (including DMN, fronto-parietal and salience networks), measured as significant changes in inter-networks connectivity parameters estimated from the temporal correlation of intrinsic functional connectivity networks.
Changes in regional brain morphometry in stress processing related areas. Measured by significant changes in regional grey matter density estimated from structural magnetic resonance imaging. | first acquisition period during 3 weeks before the intervention, second acquisition period during 3 weeks after the intervention.
Behavioural tasks: mind-wandering task | first acquisition period during 3 weeks before the intervention, second acquisition period during 3 weeks after the intervention.
  Changes in mind-wandering task, measured as changes in task-unrelated thoughts.
Changes in personality functioning. | first acquisition period during 3 weeks before the intervention, second acquisition period during 3 weeks after the intervention.
  Significant changes in levels of personality functioning measured by the operationalized psychodynamic diagnosis scale.
Experience Sampling of emotional tolerance | first acquisition period during 3 weeks before the intervention, last acquisition period during 3 weeks after the intervention. And during the intervention period everyday.
  Significant changes in self-reported capacity for emotion tolerance.
Changes in psychophysiological measurements of stress (sympathetic component) | first acquisition period during 3 weeks before the intervention, second acquisition period during 3 weeks after the intervention.
  Activation changes in psychophysiological stress parameters using Skin Conductance Response (measured as significant changes in tonic and phasic response levels) during an emotion regulation task.
Changes in psychophysiological measurements of stress (vagal component) | first acquisition period during 3 weeks before the intervention, second acquisition period during 3 weeks after the intervention.
  Activation changes in psychophysiological stress parameters using Heart Rate Variability (power analysis of high frequency sub-bands of heart rate spectrum), during an emotion regulation task.
Behavioural tasks: empathy test. | first acquisition period during 3 weeks before the intervention, second acquisition period during 3 weeks after the intervention.
  Changes in empathy test, measured as changes in levels of cognitive and affective empathy.
Changes in self-reported affective states | first acquisition period during 3 weeks before the intervention, second acquisition period during 3 weeks after the intervention.
  Significant changes in self-reported levels of negative and positive affects measured by the PANAS scale.
Changes in social functioning | first acquisition period during 3 weeks before the intervention, second acquisition period during 3 weeks after the intervention.
  Significant changes in the interpersonal competence questionnaire self-reported scale.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Dziobek, Professor, PhD., Study Chair — Humboldt Universität.
Locations (1):
- Berlin School of Mind & Brain, Humboldt Universität., Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guendelman S, Bayer M, Prehn K, Dziobek I. Towards a mechanistic understanding of mindfulness-based stress reduction (MBSR) using an RCT neuroimaging approach: Effects on regulating own stress in social and non-social situations. Neuroimage. 2022 Jul 1;254:119059. doi: 10.1016/j.neuroimage.2022.119059. Epub 2022 Mar 5. PMID 35259523
- See also: Related Info — http://www.mabstudy.de